CLINICAL TRIAL: NCT04249466
Title: Diet, Physical Activity and Glucose Tolerance in Cystic Fibrosis. Exploratory Study.
Acronym: MONA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0698
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with cystic fibrosis
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — During this consult, several parameters will be measured :
  * nutritional and physical activity parameters: Food Frequency Questionnaire (FFQ), International Physical Activity Questionnaire (IPAQ), Three-Factor Eating Questionnaire (TFEQ-R18), impedance test, anthropometric measurements, resting energy expenditure
  * demographic and clinical parameters : Family history, date of birth (month and year), sex, genotype, best forced expiratory volume (FEV) (over the 12 months preceding inclusion), bacterial colonization
  * patient treatment and biologic parameters: corticosteroid therapy (with dosage, over the 12 months preceding inclusion), antidiabetic treatment (oral or insulin), IV antibiotic treatment, corrective treatments, pancreatic enzymes, OGTT (blood glucose and insulin levels at three times), lipid balance, vitamin dosage.

SUMMARY:
Background :

Diabetes is correlated to an increase in patient morbidity and mortality. The pathophysiology of diabetes is still poorly understood. Significant variations in blood sugar have been shown over time in patients with cystic fibrosis with or without diabetes. No study has evaluated the association between the nutritional profile and the glucose tolerance in adult with cystic fibrosis, by integrating data on energy consumption (detailed nutritional profile) and energy expenditure (rest energy expenditure, body composition, and physical activity).

Given the epidemiological changes in cystic fibrosis correlated to the increased prevalence of diabetes and the clinical impact of nutritional status, the association between these factors remains to be studied.

Objectives of the study :

- Main objective :

To describe adult patients with cystic fibrosis in terms of :

* Nutritional profile
* Food behaviour
* Physical activity
* Rest energy expenditure
* Body composition - Secondary objectives : To research the association between the nutritional profile and the glucose tolerance.

DETAILED DESCRIPTION:
Study design :

The study will last 12 months. It's an observational cross-sectional study; patients are include during a scheduled review at the Cystic Fibrosis Resource and Competence Centre (CRCM de Lyon) and their participation lasts only one day. The inclusion period will last 12 months.

Expected results

The expected results are:

* Identify the inter-relationships between nutritional profile and glucose tolerance in adult patients with cystic fibrosis
* Describe the body composition and consumption on resting energy of adults with cystic fibrosis

The perspectives are:

* Propose nutritional and dietetic measures to limit the deterioration of the glucose tolerance in adult patients with cystic fibrosis
* Develop equations for evaluating consumption on resting energy specific to adult patients with cystic fibrosis in order to more specifically adapt the nutritional recommendations to each patient

The research perspectives are to compare adult patients with cystic fibrosis followed in France and Quebec in terms of:

* nutritional profiles, nutritional quality index of food and eating behaviours, resting energy expenditure, body composition
* nutritional medical practices (dietary monitoring, recommendations given to patients, intake of pancreatic enzyme).

ELIGIBILITY:
Inclusion Criteria:

* patient (male or female) with cystic fibrosis aged 18 years and over
* pancreatic insufficiency
* followed at the CRCM adult in Lyon
* patient able to understand the information given to him
* patient having previously had a medical examination during the selection visit

Exclusion Criteria:

* FEV < 30%
* lung transplant
* patient treated with insulin
* parenteral feeding on nasogastric tube or gastrostomy
* patient under guardianship or protected by law
* patient deprived of his liberty by judicial or administrative decision
* patient currently in an another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient (male or female) with cystic fibrosis or pancreatic insufficiency aged 18 years and over will answer a questionnaire to identify them in terms of:
  * Nutritional profile
  * Eating behaviour
  * Physical activity
  * Resting energy expenditure
  * Body composition
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Measurement of glycemia and insulinemia at T0, T60 and T120 min | At baseline
  Glucose tolerance is the factor studied. It's established on the basis of Oral Glucose Tolerance Test (OGTT) data, with measurement of glycemia and insulinemia at T0, T60 and T120 min.
  Carbohydrate status will be determined using the international classification:
  * Normal Glucose Tolerance (NGT) (G0 ≤ 7.0 mmol / L and G2 ≤ 7.7 mmol / L),
  * Abnormal glucose tolerance (AGT) defined by indeterminate status (INDET) (G0 ≤ 7.0 mmol / L and G2 ≤ 7.7 mmol / L, but G1 ≥ 11.1 mmol / L) or Impaired Glucose Tolerance (IGT) (G0 ≤ 7.0 mmol / L and G2> 7.7 mmol / L but <11.1 mmol / L)
  * Diabetic status (CFRD) (G0> 7.0 mmol / L or G2 ≥ 11.1 mmol / L).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de médecine interne - CRCM Lyon Adultes, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France